CLINICAL TRIAL: NCT03047876
Title: Brain Vascular Reactivity to Hypothermic Circulatory Arrest With Antegrade Cerebral Perfusion During Aortic Arch Surgery in Neonates and Infants.
Brief Title: Brain Vascular Reactivity to Hypothermic Circulatory Arrest With Antegrade Cerebral Perfusion During Aortic Arch Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 220447
Record Dates: First submitted 2017-02-03; First posted 2017-02-09 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2018-06

CONDITIONS: Cardiac; Aortic Arch Surgery; Brain Vascular; Neonates; Infants
Keywords: cardiac; aortic arch surgery; Brain vascular reactivity; neonates; infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All neonates and infants undergoing aortic arch surgery: Children, from neonatal age to late infancy, undergoing aortic arch surgery (n=20) will have cerebral perfusion measurements during surgery, including during the cooling and rewarming phase, whilst on cardiopulmonary bypass and during the recovery period in the intensive care unit
  Interventions: Procedure: aortic arch surgery

INTERVENTIONS:
Procedure: aortic arch surgery — Children, from neonatal age to late infancy, undergoing aortic arch surgery (n=20) will have cerebral perfusion measurements during surgery, including during the cooling and rewarming phase, whilst on cardiopulmonary bypass and during the recovery period in the intensive care unit

SUMMARY:
Many neonates and infants who undergo complex cardiac surgery are affected by neurological developmental delays. Whilst catastrophic events are immediately identifiable from clinical examination or by macro changes on MRI or CT scans, smaller changes are often not immediately visible or detected.

This is an observational pilot study examining brain vascular reaction to hypothermic circulatory arrest with antegrade cerebral perfusion and neuro-protection techniques during aortic arch surgery in neonates and infants. A combination of duplex ultrasound and transcranial doppler will be used to record in-depth information on the cerebrovascular changes that occur during the entire length of the surgical procedure and during the early postoperative period. The proposed techniques and equipment are non-invasive and are in use clinically to evaluate brain perfusion in a similar age group.

During aortic arch surgery, the patient's body and brain temperature is reduced to values between 18 and 24 degrees centigrade in order to decrease metabolic demand that provides a form of metabolic protection. However, there is no consensus within the clinical community regarding the optimal temperature at which to perform surgery. Moreover, in order to improve cerebral perfusion, the brain is perfused via the right internal carotid artery with cold blood. At Alder Hey Children Hospital, this surgery is undertaken by the three surgeons but, due to clinical preference, differs in relation to the temperature at which surgery is undertaken. This provides the opportunity to observe the impact of different temperatures on cerebral vascular reactivity in neonates and young infants The arguments for future comparisons and a larger randomised study will be made based on the information gained from this observational study.

DETAILED DESCRIPTION:
Children who have undergone cardiac surgery are at high risk of neurological disability. Adequate cerebral perfusion during the surgery is paramount to minimise the risk of brain injury which is a well-documented complication. Whilst this is easily identifiable through brain imaging post-operatively, less is known about intracerebral vascular reactivity that arise due to inadequate cerebral perfusion during and immediately following surgery which may result in long-term neurological deficits. Some of these changes have been observed solely through long term evaluation of childhood behaviours, as is seen in the Boston Circulatory Arrest Trial.

Aortic arch surgical repair surgery is performed in acynotic patients with conditions like Hypoplastic Aortic Arch or Interrupted Aortic Arch, or in cyanotic patients for diagnosis such as Hypoplastic Left Heart Syndrome, where a single ventricle repair is undertaken by means of a Norwood type operation.

Aortic arch surgery is performed with the aid of cardiopulmonary bypass and requires stopping the body's circulation for the time employed to repair the aortic arch. In order to provide protection to the body and to the brain, the patient's temperature is reduced to 18-25C to minimise metabolic requirements. This is particularly important for the brain so circulation can be stopped while operating on the aortic arch in a bloodless field. In recent years, techniques aimed at preserving brain perfusion during circulatory arrest have been developed. Antegrade cerebral perfusion of cold blood (18-25C) via the right internal carotid artery has been successfully employed and it is routinely used at Alder Hey Children's Hospital. Nevertheless, target brain temperature, the rate of cooling, perfusion pressure and PCO2 in arterial blood significantly influence cerebral vascular reactivity and perfusion. The optimal temperature to ensure neuroprotection is currently unknown and the temperature for cooling is based on surgeon preference rather than solid evidence.

Currently, clinical practice in the UK is to employ near infrared spectroscopy (NIRS) as an index of cerebral perfusion. Whilst this is a simple and non-invasive tool, it only measures oxygen levels in the frontal lobes, and is purely indicative of oxygenation, not absorption of oxygen by the cerebral tissue. An injured brain will continue to show normal levels of saturation on NIRS despite hypoxia (lack of oxygen) induced injury. Novel imaging techniques are now available that can provide more in-depth information on real time cerebral perfusion and quantify the magnitude of changes during and following surgery in children. One research study has employed Transcranial Doppler to monitor cerebral velocity during aortic arch surgery whilst on cardiopulmonary bypass with the aim of maintaining cerebral velocity during surgery at a level similar to before cooling. More recently, duplex ultrasound to image the cerebral vessels through the fontanelle has been employed to obtain perfusion data from both hemispheres of the brain during aortic arch surgery. Taken together, these measurement techniques provide unique novel insight into the cerebrovascular changes which occur during the surgical and post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* All neonates and infants undergoing aortic arch surgery

Exclusion Criteria:

* Procedures undertaken as an emergency
* Parents/guardians who do not wish for their child to participate
* Parents/ guardians who are unable to provide written consent

Ages: 1 Day to 1 Year | Sex: All
Age Groups: Child
Study Population: Children, from neonatal age to late infancy, undergoing aortic arch surgery (n=25) will have cerebral perfusion measurements during surgery, including during the cooling and rewarming phase, whilst on cardiopulmonary bypass and during the recovery period in the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-19 (Estimated); Study Completion 2021-03-19 (Estimated)

PRIMARY OUTCOMES:
Feasibility Data | 1 year
  Quantify the impact of surgical and post-operative clinical intervention of aortic arch surgery on cerebral perfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Alder Hey Children's Hospital, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaynor JW, Stopp C, Wypij D, Andropoulos DB, Atallah J, Atz AM, Beca J, Donofrio MT, Duncan K, Ghanayem NS, Goldberg CS, Hovels-Gurich H, Ichida F, Jacobs JP, Justo R, Latal B, Li JS, Mahle WT, McQuillen PS, Menon SC, Pemberton VL, Pike NA, Pizarro C, Shekerdemian LS, Synnes A, Williams I, Bellinger DC, Newburger JW; International Cardiac Collaborative on Neurodevelopment (ICCON) Investigators. Neurodevelopmental outcomes after cardiac surgery in infancy. Pediatrics. 2015 May;135(5):816-25. doi: 10.1542/peds.2014-3825. PMID 25917996
- [Background] McCrindle BW, Tchervenkov CI, Konstantinov IE, Williams WG, Neirotti RA, Jacobs ML, Blackstone EH; Congenital Heart Surgeons Society. Risk factors associated with mortality and interventions in 472 neonates with interrupted aortic arch: a Congenital Heart Surgeons Society study. J Thorac Cardiovasc Surg. 2005 Feb;129(2):343-50. doi: 10.1016/j.jtcvs.2004.10.004. PMID 15678045
- [Background] Wypij D, Newburger JW, Rappaport LA, duPlessis AJ, Jonas RA, Wernovsky G, Lin M, Bellinger DC. The effect of duration of deep hypothermic circulatory arrest in infant heart surgery on late neurodevelopment: the Boston Circulatory Arrest Trial. J Thorac Cardiovasc Surg. 2003 Nov;126(5):1397-403. doi: 10.1016/s0022-5223(03)00940-1. PMID 14666011
- [Background] Andropoulos DB, Stayer SA, McKenzie ED, Fraser CD Jr. Regional low-flow perfusion provides comparable blood flow and oxygenation to both cerebral hemispheres during neonatal aortic arch reconstruction. J Thorac Cardiovasc Surg. 2003 Dec;126(6):1712-7. doi: 10.1016/s0022-5223(03)01027-4. PMID 14688677
- [Background] Ruffer A, Tischer P, Munch F, Purbojo A, Toka O, Rascher W, Cesnjevar RA, Jungert J. Comparable Cerebral Blood Flow in Both Hemispheres During Regional Cerebral Perfusion in Infant Aortic Arch Surgery. Ann Thorac Surg. 2017 Jan;103(1):178-185. doi: 10.1016/j.athoracsur.2016.05.088. Epub 2016 Aug 23. PMID 27526653